CLINICAL TRIAL: NCT06544642
Title: A Phase 1 Combined Single and Multiple Ascending Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Food Effect and Biomarker Response of ASP5502 in Healthy Adults and Participants With Primary Sjögren's Syndrome
Brief Title: A Study to Evaluate the Effects of ASP5502 in Healthy Adults and Adults With Primary Sjögren's Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 5502-CL-0001
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers; Sjögren's Syndrome
Keywords: ASP5502; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; Food Effect
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 - Single Ascending Dose in Healthy participants (Dose Escalation Cohort) (Experimental): Participants will receive a single oral dose of ASP5502 or Placebo on Day 1.
  Interventions: Drug: ASP5502; Drug: Placebo
- Part 1 - Single Ascending Dose in Healthy participants (Food Effect Cohort) (Experimental): Participants will receive a single oral dose of ASP5502 or Placebo under fasting conditions on period 1 Day 1 and single dose of ASP5502 or Placebo under fed conditions on period 2 Day 1.
  Interventions: Drug: ASP5502; Drug: Placebo
- Part 2 - Multiple Ascending Dose in Healthy participants (Experimental): Participants will receive daily oral doses of ASP5502 or placebo for 14 days.
  Interventions: Drug: ASP5502; Drug: Placebo
- Part 3 - Repeated Dose in Participants with pSS (Experimental): Participants will receive daily oral doses of ASP5502 for 28 days.
  Interventions: Drug: ASP5502

INTERVENTIONS:
Drug: ASP5502 — Oral
Drug: Placebo — Oral
  Arms: Part 1 - Single Ascending Dose in Healthy participants (Dose Escalation Cohort); Part 1 - Single Ascending Dose in Healthy participants (Food Effect Cohort); Part 2 - Multiple Ascending Dose in Healthy participants

SUMMARY:
Primary Sjögren's syndrome (pSS) is a condition when the body's immune system attacks glands that produce fluids, such as the tear and saliva glands. This leads to dry eyes and a dry mouth. However, other symptoms may occur such as fatigue, joint pain, and skin problems. These symptoms can be severe. Symptoms can be treated but there is an unmet need to treat the actual condition.

In this study, ASP5502 is being given to humans for the first time. The people taking part are healthy adults or adults with pSS. The main aims of the study are to check the safety of ASP5502 and how people tolerate ASP5502.

This study will be in 3 parts. In Part 1, healthy men and women will take tablets of ASP5502 or a placebo just once. In this study, the placebo looks like the ASP5502 tablet but doesn't have any medicine in it. Different small groups of people will take a lower to a higher dose of ASP5502 or a placebo. This will happen one group after another. One small group will take tablets of ASP5502 or placebo with and without food. This is to find out if food affects how the body processes ASP5502.

After their dose, people will stay in the medical center for a few nights. This is to have blood tests, electrocardiograms (ECGs) to check heart health, and other safety checks, and to report any medical problems. One of these checks is to have their heart continuously tracked during the first night. This is called telemetry. People who take tablets of ASP5502 or placebo with and without food will stay in the medical center for a few extra nights.

In Part 2, healthy men and women will take tablets of ASP5502 or a placebo. They will do this once a day for 2 weeks (14 days). Different small groups of people will take a lower to a higher dose of ASP5502 or a placebo. This will happen one group after another.

After taking ASP5502 or the placebo, people will stay in the medical center for a few nights. This is to have blood tests, ECGs to check heart health, and other safety checks, and to report any medical problems. Telemetry will also be done continuously during the first night.

In Part 3, men and women with pSS will take tablets of ASP5502. They will do this once a day for 4 weeks (28 days). Different small groups of people will take a lower to a higher dose of ASP5502. This will either happen for one group after another, or just for 1 group. The number of groups and the doses taken will be worked out from the results from Part 1 and Part 2 of this study. People will stay in the medical center for a couple of nights. This will happen for their first dose, then again after about 2 weeks and 4 weeks of treatment. As in Parts 1 and 2, this is to have blood tests, ECGs to check heart health, and other safety checks, and to report any medical problems.

In all parts of the study, people will return to the medical center about 1 week after their final blood sample is taken, for health check. People in parts 2 and 3 will also receive a telephone call safety check about 4 weeks after their last dose of ASP5502.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Healthy Participants

* Participant is healthy and has no clinically significant medical conditions based on the review of the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -2 or day -1.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a women of childbearing potential (WOCBP)
  * WOCBP who has a negative blood pregnancy test at screening and a urine pregnancy test on day -2 and agrees to follow the contraceptive guidance from the time of informed consent through at least 5 half-lives or 30 days, whichever is longer, after final study intervention administration. Female participants on hormonal contraceptives must also be using a double barrier method as defined in Contraceptive Requirements.
* Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Female participant must not donate ova starting at first administration of study intervention and throughout the investigational period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Male participant must not donate sperm during the treatment period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Participant agrees not to participate in another interventional study while participating in the present study from the time of signing informed consent through the end of study visit.
* Participant has a body mass index (BMI) range of 18.5 to 30.0 kg/m^2 inclusive and weighs at least 50 kg for male and 40 kg for female at screening.

Inclusion Criteria for Participants with pSS

* Participant is diagnosed based on the 2016 American College of Rheumatology (ACR)- European Alliance of Associations for Rheumatology (EULAR) Classification Criteria for pSS. Diagnosis should have been established at least 6 months prior to day -1 and no clinically significant medical condition is present on the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -1.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a WOCBP
  * WOCBP who has a negative blood pregnancy test at screening and a urine pregnancy test on day -1 and agrees to follow the contraceptive guidance from the time of informed consent through at least 5 half-lives or 30 days, whichever is longer, after final study intervention administration. Female participants on hormonal contraceptives are allowed ONLY if the participant also agrees to use a double barrier method (condom and spermicide) and the results from the 4β hydroxycholesterol assessment in Part 2 are negative.
  * WOCBP must also be using a double barrier method as defined in Contraceptive Requirements.
* Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Female participant must not donate ova starting at first administration of study intervention and throughout the investigational period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Male participant must not donate sperm during the treatment period and for 5 half-lives or 30 days, whichever is longer, after final study intervention administration.
* Participant agrees not to participate in another interventional study while participating in the present study from the time of signing informed consent through the end of study visit.
* Participant has a BMI range of 18.5 to 30.0 kg/m^2 inclusive and weighs at least 50 kg for male and 40 kg for female at screening.

Exclusion Criteria:

Exclusion Criteria for Healthy Participants

* Participant has been pregnant within 6 months prior to screening.
* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has a history of malignancy within 2 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that is considered cured with minimal risk of recurrence).
* Participant has had major surgery (e.g., requiring general anesthesia) within 90 days before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study or within 5 half-lives after the last dose of study intervention administration or end of study visit, whichever is longer.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 28 days prior to day -1.
* Participant has a positive QuantiFERON®-TB Gold test at screening.
* Participant has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) criteria within 2 years before screening.
* Participant has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, a family history of long QT syndrome or taking any QT prolonging medication.
* Participant has used any prescribed or nonprescribed drugs (including vitamins and natural and herbal remedies, e.g., St. John's Wort) in the 28 days prior to study intervention administration, except for contraceptive use, hormone replacement therapy (HRT) use and occasional use of acetaminophen (up to 2 g/day).
* Participant has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Participant has received a vaccine within the 2 weeks prior to day -1 or will have a vaccine dose before the follow-up visit.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any of the liver safety monitoring panel (alkaline phosphatase [ALP], alanine transaminase [ALT], aspartate aminotransferase [AST] and total bilirubin [TBL]) above the upper limit of normal (ULN) on day -2. In such a case, the assessment may be repeated once.
* Participant has creatinine level outside normal limits on day -2. In such a case, the assessment may be repeated once.
* Participant has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -2. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean corrected QT interval using Fridericia's correction formula (QTcF) of > 430 msec (for male participants) and > 450 msec (for female participants) on day -2. If the mean QTcF exceeds these limits, 1 additional triplicate ECG may be taken.
* Participant tests positive for alcohol at screening or on day -2.
* Participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine and opiates) at screening or on day -2.
* Participant tests positive for cannabinoids on day -2.
* Participant has a positive rapid coronavirus disease (COVID) antigen test on day -2.
* Participant has a positive serology test for hepatitis A virus (HAV) antibodies (immunoglobulin M [IgM]), hemoglobin C (HBc) antibodies, hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV) antibodies or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP5502 or comparator or any components of the formulation used.
* Participant has smoked, used tobacco-containing products or nicotine or nicotine-containing products (e.g., electronic vapes) within 6 months prior to screening or the participant tests positive for cotinine at screening or day -2.
* Participant has a history of consuming > 10 units for male or > 8 units for female participants of alcoholic beverages per week within 3 months prior to screening (note: 1 unit = 12 ounces of beer, 5 ounces of wine, 1.5 ounce of spirits/hard liquor).
* Participant has used any drugs of abuse (e.g., amphetamines, barbiturates, benzodiazepines, cocaine and/or opiates) within 3 months prior to day -1.
* Participant has had significant blood loss, donated >/= 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Participant has had previous exposure with ASP5502.
* Participant is an employee of Astellas, the study-related clinical research organizations (CROs) or the clinical unit.

Exclusion Criteria for Participants with pSS

* Participant has been diagnosed with secondary Sjögren's syndrome or any other systemic autoimmune disease (e.g. rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis).
* Participant has severe complications of Sjögren's syndrome, such as neurologic or cardiac involvement, interstitial lung disease and severe myositis.
* Participant is using immunosuppressant therapy (e.g., methotrexate, azathioprine, mycophenolate mofetil), B-cell depleting agents (e.g., rituximab, belimimab), Janus kinase inhibitors (JAKi) (e.g., tofacitinib), calcineurin inhibitors (e.g., tacrolimus, cyclosporin), and other biologics (e.g., abatacept, cyclophosphamide, leflunomide).
* Participant receives corticosteroid therapy exceeding 10 mg prednisone equivalents per day.
* Participant has been pregnant within 6 months prior to screening.
* Participant has any history or evidence of any not-related to pSS clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has a history of malignancy within 2 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that is considered cured with minimal risk of recurrence).
* Participant has had major surgery (e.g., requiring general anesthesia) within 90 days before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study or within 5 half-lives after the last dose of study intervention administration or end of study visit, whichever is longer.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 28 days prior to day -1.
* Participant has a past history of serious opportunistic infections.
* Participant has a positive QuantiFERON®-TB Gold test at screening.
* Participant has a positive rapid COVID antigen test on day -1.
* Participant has a history of drug or alcohol abuse according to DSM-5 criteria within 2 years before screening.
* Participant has any of the liver safety monitoring panel (ALP, ALT, AST and TBL) above the ULN on day -1. In such a case, the assessment may be repeated once.
* Participant has creatinine level outside normal limits on day -1. In such a case, the assessment may be repeated once.
* Participant has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean corrected QTcF of > 450 msec on day -1.
* Participant has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease or a family history of long QT syndrome.
* Participant is using QT prolongating medication such as antiarrhythmics (e.g. amiodarone, sotalol, ibutilide, dofitilide, disopyramide), antipsychotic (e.g. chlorpromazine, haloperidol), antidepressants (e.g. citalopram), antibiotics (e.g. sparfloxacin, ciprofloxacin, erythromycin, azithromycin, clarithromycin) or antiemetics (e.g. domperidone).
* Participant has used any Cytochrome P450 (CYP) 3A4 inducer of metabolism (e.g., barbiturates and phenytoin, barbiturates, carbamazepine, bosentan, felbamate, griseofulvin, oxcarbazepine, rifampicin, topiramate, rifabutin, rufinamide, aprepitant and products containing St. John's wort) or HIV protease inhibitors, HCV protease inhibitor or non-nucleoside reverse transcriptase inhibitors (e.g., nelfinavir, ritonavir, darunavir/ritonavir, (fos)amprenavir/ritonavir, lopinavir/ritonavir, tipranavir/ritonavir, boceprevir, telaprevir and nevirapine) within 3 months prior to day -1.
* Participant has used any narrow therapeutic index CYP3A4 substrate (e.g., alfentanil, cyclosporine, dihydroergotamine, ergotamine, everolimus, fentanyl, pimozide, quinidine, sirolimus, and tacrolimus) within 24 hours prior to day -1.
* Participant has received a vaccine within the 2 weeks prior to first study intervention administration or will have a vaccine dose before the follow-up visit.
* Present or previous history of participation in a study of the study intervention.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP5502 or any components of the formulation used.
* Participant is an employee of Astellas, the study-related clinical research organizations (CROs) or the clinical unit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to Day 58
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
Number of participants with laboratory value abnormalities and/or AEs | Up to Day 38
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to Day 38
  Number of participants with potentially clinically significant vital sign values.
Number of participants with 12-lead ECG abnormalities and/or AEs | Up to Day 38
  Number of participants with potentially clinically significant 12-lead ECG values.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP5502 in plasma: maximum concentration (Cmax) | Up to Day 29
  Cmax will be recorded from the PK plasma samples collected.
PK of ASP5502 in plasma: area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast) [Part 1] | Up to Day 7
  AUClast will be recorded from the PK plasma samples collected.
PK of ASP5502 in plasma: area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf) [Part 1] | Up to Day 7
  AUCinf will be recorded from the PK plasma samples collected.
PK of ASP5502 in plasma: area under the concentration-time curve from time of dosing to 24 hours post dose (AUC24) [Part 2 & Part 3] | Up to Day 2
  AUC24 will be recorded from the PK plasma samples collected.
PK of ASP5502 in plasma: area under the concentration-time curve during a dosing interval, where tau is the length of the dosing interval (AUCtau) [Part 2 & Part 3] | Up to Day 29
  AUCtau will be recorded from the PK plasma samples collected.
PK of ASP5502 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) [Part 2 & Part 3] | Up to Day 29
  Ctrough will be recorded from the PK plasma samples collected.
Change from baseline in concentration-QT [Part 1 & Part 2] | Baseline up to Day 20
  QT will be measured using ECG machine at site. Concentration will be recorded from PK plasma sample.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Fortrea Clinical Research Unit Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.